CLINICAL TRIAL: NCT02619968
Title: Effectiveness of Physical Exercise With Flow Restriction on the Diameter and the Flow of the Blood Vessels of the Forearm in Chronic Kidney Disease: a Randomized Clinical Trial
Brief Title: Physical Exercise With Flow Restriction of the Forearm in Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Jefferson Belarmino Nunes Barbosa, postgraduate in integrated multidisciplinary residency in health, concentration area in physical therapy in nephrology, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 07587234403
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic renal failure; Arteriovenous fistula; Isometric exercises; Vascular endothelium
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental group (Experimental): Will be held isometric and isotonic concentric to the flexor muscles of the elbow and wrist using tennis ball, halter and handgrip added to partial occlusion of blood flow to tourniquet application.
  Application of the tourniquet Will be held in conjunction with exercises for the experimental group.
  Tennis ball: will initially be 3 sets, where one series with 10 grips, increasing 5 grips every week, 60 seconds rest every series.
  Halter: are performed with load of 1 kg, 2 kg and 3 kg. Handgrip: they will be performed 3 sets of dynamic manual hold exercises in the intensity of 40% of MVC.
  Home program: at home will be performed isometric exercises with tennis ball on the same frequency as in performing ambulatory without applying the tensiometer.
  Interventions: Other: experimental group
- Group control (Sham Comparator): Will be held the same isometric and isotonic concentric ambulatory and home with the same duration, frequency and intensity, except is not to apply the tourniquet.
  Interventions: Other: experimental group

INTERVENTIONS:
Other: experimental group — Will be held isometric and isotonic concentric to the flexor muscles of the elbow and wrist using tennis ball, halter and handgrip added to partial occlusion of blood flow to tourniquet application. The Application of the tourniquet will be held in conjunction with exercises for the experimental group.

SUMMARY:
The aim of this study is to analyze the effectiveness of physical exercise with blood flow restriction on the diameter and the flow of vessels, muscle strength and circumference of the forearm in patients with CKD prior to making FAV.

DETAILED DESCRIPTION:
Definitions of goals

General Analyze the effectiveness of physical exercise with blood flow restriction on the diameter and the flow of vessels, muscle strength and circumference of the forearm in patients with CKD prior to making arteriovenous fistula.

Specific

* Draw the profile of patients with CKD as the clinical and laboratory features (hematocrit, hemoglobin, urea, creatinine) and glomerular filtration rate;
* Assess the vascular conditions, muscle strength and circumference of the upper limb of the non-dominant forearm before and after exercise programs;
* Compare the physical exercise programs with and without blood flow restriction vascular changes, muscle strength and circumference of the non-dominant arm;
* To correlate the diameter measurements and blood flow to the muscle strength and circumference of the upper limb not dominant.

Methodology Study design This is a randomized controlled trial, blind and endowed with allocation concealment to be developed in Physiotherapy clinic and Nephrology at the Clinical Hospital, Federal University of Pernambuco and Cardiopulmonary Physiotherapy Laboratory in the Department of Physical Therapy, Federal University of Pernambuco, the From December 2015 to November 2016, following approval of the Committee of Ethics in Research / the Health Sciences Center.

After approval by Committee of Ethics in Research / the Health Sciences Center according to Resolution 466/2012 of the National Health Council and the explanation of the study, participants will be asked to sign the Informed Consent (IC).

The recruitment and evaluations will be carried out by a single evaluator, who will be blinded when randomization, allocation and interventions.

Inclusion criteria The sample will consist of patients with Chronic Kidney Disease (CKD) Stage 4 or 5, of both sexes, from 18 years of age, in conservative or dialysis treatment with medical indication of arteriovenous fistula as an achievement of hemodialysis.

Exclusion criteria Are excluded those that present cognitive impairment or changes that hinder understanding, realization of activities and interpretation of the issues; a history of making arteriovenous fistula in both upper limbs or some other type of vascular surgery in upper limbs, with some type of vascular access in upper limbs or in nearby regions; to develop some kind of manual work with heavy loads; Trauma-orthopedic lesions in the cervical, shoulder, elbow, wrist and untreated (or) hand; signs of thrombophlebitis and hypoplasia / agenesis of the upper limbs.

Study design After enrollment in the nephrology clinic of the Clinical Hospital / Federal University of Pernambuco will initially applied the Mini-Mental State Examination (MMSE), to exclude the possibility of cognitive impairment.

Anamnesis It will be performed in the clinic of Nephrology, after the MMSE through questionnaire with open and closed questions. The data used are: sex, age (years), weight (kg), height (m), body mass index (BMI), blood pressure (BP) (mmHg) (Brazilian Society of Cardiology, 2010), etiology and stage CKD, serum creatinine (mg / dL) and urea (mg / dL) of the last test reported in medical records and Glomerular Filtration Rate (mL / min) (Cockcroft; GAULT, 1976), hematocrit (%) and hemoglobin (g / dL) and current medications. These data will be checked in an interview and medical records of patients that will be opened during the interview will last approximately 15 minutes. After the date for physical examination will be scheduled.

Physical exam It will be held on Cardiopulmonary Physiotherapy laboratory at Federal University of Pernambuco. The patient will designate its upper limb non-domimant, according to the guidelines of the Kidney Disease Outcomes Quality Initiative Guidelines (VASCULAR ACCESS WORK GROUP, 2006). Then will take place the forearm circumference assessments, morphology of the vessels and handgrip strength. This will take the total duration of approximately 50 minutes.

Circumference forearm The circumference of the forearm will be performed by perimetry (tape nylon). The patient will be sitting in the chair with the supinated forearm and elbow flexed at 90 °. The tape is positioned at the distal 2 cm of the cubital fossa (KONG et al, 2014). Will be held 3 measurements, registering the highest value.

Morphology vessel To evaluate the radial artery are measured the internal cross-sectional diameter (mm) at flow rate of [systolic peak (cm / sec) and average velocity (cm / s)]. For the cephalic vein, will be measured basal venous outside diameter (mm) and venous outer diameter after placement of tourniquet (mm), and distensibility of the cephalic vein (%) for upper limb (UL) by ultrasonography [Sonoace R3 ( Samsung Medison - South Korea)]. A linear transducer 10 megahertz multifrequency (RUS et al, 2005; Kumar et al, 2010; RUS et al, 2005) will be used.

Handgrip strength Will be assessed by manual dynamometer (Smedley Dynamometer - Type hand mark Saehan - Korea) to evaluate the maximum voluntary contraction (MVC). Will be conducted two tests with rest interval of five minutes after the first reading, is considered the greatest value.

Evaluations of the circumference of the forearm, the vessel morphology and handgrip strength will be performed by the same evaluator before and after the interventions, which will be blinded as to the randomization of patients to interventions and their implementation (KONG et al, 2014).

Intervention Protocol Will run for eight weeks for each patient, being developed in five days of the week (2 days with supervision by the physiotherapist on an outpatient basis and 3 days at home).

After randomization, patients will be divided into two groups, experimental (EG) and control (CG).

Experimental group For experimental group, will be held isometric and isotonic concentric to the flexor muscles of the elbow and wrist using tennis ball, halter and handgrip added to partial occlusion of blood flow to tourniquet application.

Between exercise modalities will be given two minutes apart.

Partial occlusion protocol for prescription tourniquet for treatment:

Application of the tourniquet Will be held in conjunction with exercises for the experimental group group will be determined in the interview. The partial occlusion of blood flow will be induced by inflation of a tensiometer on the upper arm and the stethoscope is placed on the medial aspect of the elbow crease, (3M ™ Littmann® Classic II SE, USA) to verify the absence of the arterial pulse. After the disappearance of the sound, the cuff is deflated slowly, observing the first arterial pulse, which is used 50% of it to occlusion during training, and graduated in mmHg. This pressure will be maintained for the three types of exercises in all grades, including the 2-minute interval during periods of rest (LOENNEKE et al, 2015).

Tennis ball For exercises with tennis ball, will initially be 3 sets, where one series with 10 grips (each squeeze lasting 3 seconds, 1 second rest), increasing 5 grips every week, 60 seconds rest every series. There will be two minutes of rest, then will repeat the same sequence. After, it will be given two minutes of rest for the next activity (KONG et al, 2014).

Halter The exercises are performed with load of 1 kg (during the first two weeks of training), 2 kg (for the last two weeks of the first month) and 3 kg for the last 4 weeks. The exercise will be conducted through elbow flexion, with the patient seated. The exercise will consist of three sets of 10 movements, maintaining shrinkage for 3 seconds, followed by 1-second standing (extension member). Between each series of 10 contractions will rest 60 seconds. 2 will be given minutes of rest at the end of this, before the next activity (SALIMI et al, 2013).

Handgrip They will be performed 3 sets of dynamic manual hold exercises in the intensity of 40% of MVC, with a frequency of 20 contractions per minute (duty cycle of 2/2 of contraction and 1 second rest). After 3 sets of 20 contractions, will be given one minute of rest. This activity will be performed to volitional fatigue, and recorded the time and amount of sets performed per patient (Hunt et al, 2012; UY et al, 2013).

Home program At home will be performed isometric exercises with tennis ball on the same frequency as in performing ambulatory without applying the tensiometer. Will be held the two sequences (3 sets of 10 grips) once daily for three days this week, which will be guided verbally by the trainer and delivered all the guidelines through leaflet, materials for the exercise and a daily control conducting training. Links will be held daily to help control procedures. Appendix 6 presents the check-list for muscle training the experimental group (Hunt et al, 2012).

Group control In the control group (CG) will be held the same isometric and isotonic concentric ambulatory and home with the same duration, frequency and intensity, except is not to apply the tourniquet.

Completion of the program The program will end at the end of the 3rd day of the last week of the completion of home procedures, and scheduled the revaluation and its realization in sequence.

It will be recorded the frequency of patients to outpatient care and conducting training at home in both groups by the instructor. Patients who do not carry 75% of the program will be given as loss of tracking.

Tabulation plan and analysis Spreadsheets Data will be recorded primarily in chips assessments of each patient, and then will be transferred to the Microsoft Office Excel spreadsheets type, version 2010® and later to the software Statistical Package for the Social Sciences (SPSS) version 20.0 for Windows for statistical analysis.

Statistical methods for data analysis Initially descriptive data analysis will be carried out, which may be presented as mean ± standard deviation, confidence interval of 95% and frequency distribution. The normal distribution is used for the continuous variables, using the Shapiro-Wilk test and the homogeneity using Levene's test. At the end of the program will be realized the Student t test for paired comparing pre and post between the same groups and the Mann-Whitney test for comparisons between groups of non-paired samples. For correlations will be used the Pearson or Spearman correlation test. It will be considered p value less than 0.05 as significant. For data analysis, SPSS for Windows version 20.0 is used.

Budget - funding

Material - Cost (R $) A4 reams of paper, 75g / m² - 5 units - 50.00 Black ink cartridges for the printer - 03 units - 90.00 Color ink cartridges for printer - 02 units - 70.00 Pens - 01 box with 50 units. - 8:00 pm Test copies and instruments - 35.00 Clipboard - 7.00 Photo copies - 50.00 1 compact disk box with 10 units - 10.00 Aneroid sphygmomanometer manual Premium - 1 unit - 60.00 Handgrip with adjustable load of 5 to 20 kg - 3 units (42,00 each R $) - 126.00 Handgrip with adjustable load of 10 to 40 kg - 3 units (55,00 each R $) - 165.00 Rubberized dumbbells 1 kg - 3 units (R $ 12.90 each) - 38.70 Rubberized dumbbells 2 kg - 3 units (R $ 20.90 each) - 62.70 Rubberized dumbbells 3 kg - 3 units (R $ 29.90 each) -89.70 Tennis Balls - 54 units (R $ 6.00 each) - 324.00 Nylon tape metric - 1 unit - 5.00 Ultrasound R3 Sonoace (Samsung Medison - South Korea) * - 75,000.00 Stethoscope 3M ™ Littmann Classic II SE, USA - 420.00 Manual dynamometer (Smedley Dinamometer - Type hand mark Saehan - Korea * - 1,499.00 Total - 78122.10

* Available in the research sites. The total cost for the research project will be the responsibility of the researcher, at no cost to the institution.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Chronic Kidney Disease (CKD) stage 4 or 5;
* In conservative or dialysis treatment;
* Medical indication of arteriovenous fistula as an achievement of HD.

Exclusion Criteria:

* Cognitive impairment or changes that hinder understanding, realization of activities and interpretation of the issues;
* a history of making FAV in both upper limbs or some other type of vascular surgery in upper limbs, with some type of vascular access in upper limbs or in nearby regions;
* to develop some kind of manual work with heavy loads;
* Trauma-orthopedic lesions in the cervical, shoulder, elbow, wrist and untreated (or) hand;
* Signs of thrombophlebitis and hypoplasia / agenesis of the upper limbs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Increasing the diameter of the cephalic vein | 8 weeks of training for each patient
  Increasing the diameter of the cephalic vein of at least 0.22 mm

SECONDARY OUTCOMES:
Increasing the diameter of the radial artery | 8 weeks of training for each patient
Radial artery blood flow | 8 weeks of training for each patient
Forearm Circumference | 8 weeks of training for each patient
Muscle strength of the forearm | 8 weeks of training for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson B Barbosa, physiotherapist, Principal Investigator — Universidade Federal de Pernambuco

REFERENCES:
- [Background] Levey AS, Coresh J. Chronic kidney disease. Lancet. 2012 Jan 14;379(9811):165-80. doi: 10.1016/S0140-6736(11)60178-5. Epub 2011 Aug 15. PMID 21840587
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Lugon JR. End-stage renal disease and chronic kidney disease in Brazil. Ethn Dis. 2009 Spring;19(1 Suppl 1):S1-7-9. PMID 19484865
- [Background] Rus RR, Ponikvar R, Kenda RB, Buturovic-Ponikvar J. Effect of local physical training on the forearm arteries and veins in patients with end-stage renal disease. Blood Purif. 2003;21(6):389-94. doi: 10.1159/000073441. PMID 14586181
- [Background] Rus RR, Ponikvar R, Kenda RB, Buturovic-Ponikvar J. Effect of intermittent compression of upper arm veins on forearm vessels in patients with end-stage renal disease. Hemodial Int. 2005 Jul;9(3):275-80. doi: 10.1111/j.1492-7535.2005.01142.x. PMID 16191078
- [Background] Kumar S, Seward J, Wilcox A, Torella F. Influence of muscle training on resting blood flow and forearm vessel diameter in patients with chronic renal failure. Br J Surg. 2010 Jun;97(6):835-8. doi: 10.1002/bjs.7004. PMID 20309951
- [Derived] Nantakool S, Reanpang T, Prasannarong M, Pongtam S, Rerkasem K. Upper limb exercise for arteriovenous fistula maturation in people requiring permanent haemodialysis access. Cochrane Database Syst Rev. 2022 Oct 3;10(10):CD013327. doi: 10.1002/14651858.CD013327.pub2. PMID 36184076